CLINICAL TRIAL: NCT07376122
Title: A Prospective, Single-Arm Pilot Study Evaluating the Effect of Robotic Spinal Mobilization (BackHug) on Mobility, Pain, and Sleep in Parkinson's Disease
Brief Title: Pilot Study of Robotic Spinal Mobilization in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacla Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM-PD-2026-01
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD)
Keywords: Axial Rigidity, Spinal Mobilization, Robotic Therapy, Chronic Pain, Sleep Quality, Gait Disorders
MeSH Terms: conditions — Parkinson Disease; Chronic Pain; Sleep Initiation and Maintenance Disorders; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: BackHug Robotic Therapy (Experimental)
  Interventions: Device: BackHug Robotic Spinal Mobilization System

INTERVENTIONS:
Device: BackHug Robotic Spinal Mobilization System — Participants will receive spinal mobilization therapy using the BackHug Robotic System. The device comprises a treatment bed with 26 robotic therapeutic heads ('fingers') that deliver targeted mechanical pressure to the paraspinal muscles and intervertebral joints of the cervical, thoracic, and lumbar spine. The mechanism is designed to mobilize stiff spinal segments and reduce paraspinal muscle tension (axial rigidity).
  Protocol:
  Regimen: Four (4) sessions administered over a two-week period.
  Duration: 40 minutes per session.
  Personalization: Treatment intensity and speed are adjusted to individual user tolerance via the device's control app, while maintaining a standardized focus on the full spine.
  Mechanism: Real-time load sensing adapts pressure to the user's specific spinal curvature.

SUMMARY:
This interventional pilot study will evaluate the safety and clinical efficacy of robotic spinal mobilization in community-dwelling adults with Parkinson's Disease (PD). The primary objective is to determine if the mechanical release of axial rigidity using the BackHug device correlates with measurable improvements in functional mobility and postural stability.

Participants will be prospectively recruited and assigned to receive a standardized course of robotic therapy. The intervention consists of a series of 40-minute sessions administered over a defined observation period. The device features 26 robotic therapeutic heads designed to deliver targeted deep-tissue mobilization to the paraspinal muscles and intervertebral joints of the thoracic and lumbar spine.

Key outcomes will be assessed using a repeated-measures design. Functional mobility (3-Meter Timed Up and Go) and functional strength (30-Second Sit-to-Stand) will be measured immediately before and after specific sessions to quantify acute therapeutic effects. Additionally, subjective metrics for chronic back pain (VAS) and sleep quality will be monitored to assess longitudinal benefits. This study aims to validate non-invasive mechanical mobilization as a scalable adjunct therapy for managing the 'axial' symptoms of Parkinson's Disease.

DETAILED DESCRIPTION:
Study Rationale: Axial rigidity is a cardinal motor feature of Parkinson's Disease (PD), characterized by stiffness in the trunk and spine. This symptom contributes significantly to gait impairment, balance dysfunction, and chronic pain, yet often shows limited response to standard dopaminergic medication. This interventional study will investigate the utility of the BackHug robotic device to mechanically mobilize the thoracic and lumbar spine, evaluating the hypothesis that reducing axial stiffness improves systemic mobility.

Study Design: This is a prospective, single-arm, open-label interventional pilot study.

The Intervention (BackHug): Participants will be assigned to receive therapy on the BackHug device.

Duration: 40 minutes per session.

Mechanism: 26 robotic fingers delivering targeted pressure to the paraspinal muscles.

Settings: Intensity and speed will be personalized to user tolerance but standardized to target the neck, shoulders, and full back.

Eligibility Criteria:

Inclusion: Adults (18-75) with confirmed PD; Hoehn and Yahr Stages 1-3; Ability to walk independently for 5 minutes.

Exclusion: Serious bone pathology (malignancy, infection, severe osteoporosis/osteomalacia); Inflammatory arthritides; Non-PD neurological conditions (spinal cord compression); Vascular risks (aortic aneurysm).

Study Protocol:

Screening & Baseline: Candidates will undergo safety screening against contraindications. Baseline functional metrics (TUG, STS) and subjective scores (VAS, Sleep) will be recorded.

Intervention Phase:

Pre-Therapy Testing: Functional tests performed immediately prior to therapy.

Therapy Administration: Automated robotic mobilization session.

Post-Therapy Testing: Functional tests repeated immediately post-session to capture acute motor changes.

Follow-up: Final assessments will be conducted at the end of the protocol to evaluate short-term retention of benefits.

Outcome Measures:

Primary: Change in Functional Mobility via 3-Meter Timed Up and Go (TUG).

Secondary: Change in Functional Strength via 30-Second Sit-to-Stand (STS); Change in Pain Intensity via VAS (0-10); Change in Sleep Quality via Likert Scale.

Exploratory: Proprioception and fine motor control (Finger-Nose, Toe Tapping).

Quality Assurance & Data Management Plan:

Data Validation: All functional assessments will be administered by trained clinical staff using standardized protocols to ensure inter-rater reliability.

Source Data Verification: Primary data will be recorded on source documents (Case Report Forms). Where consent is granted, video recordings of functional tests will serve as source data for timing verification.

Data Checks: The electronic database will employ logic checks (e.g., range limits for Age and VAS scores) to prevent data entry errors.

Missing Data Plan: The study will utilize a Last Observation Carried Forward (LOCF) approach for minor missing data points, or conduct analysis on a Per-Protocol basis for the primary endpoint.

Statistical Analysis Plan:

Sample Size: The study aims to recruit a cohort sufficient to generate effect size estimates for a future randomized controlled trial.

Analysis: Paired t-tests (or Wilcoxon signed-rank tests for non-parametric data) will be used to compare Pre- vs. Post-intervention scores. Descriptive statistics will summarize demographic baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Participants must have a confirmed clinical diagnosis of Parkinson's Disease.
* Disease Severity: Hoehn and Yahr Scale Stage 3 or below (indicating mild to moderate disability; capable of independent balance).
* Functional Mobility: Ability to walk independently for approximately 5 minutes. Use of walking poles is permitted; however, reliance on a walking frame (Zimmer frame) or wheelchair excludes participation.
* Age: 18 to 80 years.

Exclusion Criteria:

Participants are excluded if they present with any absolute contraindication to mechanical spinal mobilization, including:

* Spinal Pathology & Trauma: History of spinal malignancy (benign or malignant tumors), active spinal infection (e.g., tuberculosis), severe congenital defects (dysplasia), or currently healing spinal fractures/dislocations.
* Metabolic & Inflammatory Bone Disease: Diagnosed severe Osteomalacia or severe Rheumatoid Arthritis (due to ligamentous instability risk).
* Neurological Contraindications (Non-PD): Evidence of spinal cord compression, Cauda Equina syndrome, or other serious neurological conditions causing spinal instability or loss of sensation.
* Vascular & Hematological Risks: History of aortic dysfunction (e.g., abdominal aortic aneurysm), severe haemophilia, or unmanaged coagulation disorders causing bleeding into joints.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Mobility (Gait Speed and Agility) | Baseline and 4 weeks.
  Functional mobility is assessed using the Timed Up and Go (TUG) Test (or a similar timed walking task). Participants are timed (in seconds) as they rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. A shorter time indicates better mobility and reduced bradykinesia.

SECONDARY OUTCOMES:
Change in Subjective Back Pain Intensity | Baseline and 4 weeks.
  Participants self-report their current level of back pain or discomfort using the Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst possible pain.
Change in Self-Reported Sleep Quality | Baseline and 4 weeks.
  Participants rate their overall quality of sleep using a 5-point Likert scale. The scale ranges from 0 to 5, where:
  5 = Very Poor (Frequent waking, discomfort)
  0 = Excellent (Uninterrupted, restful sleep) Higher scores indicate an improvement in sleep quality.
Change in Functional Lower Limb Strength (30-Second Sit-to-Stand Test)' | Baseline (Session 1) and Post-Intervention (Session 4, approximately 2 weeks later)
  Participants are instructed to sit in a chair with arms crossed over their chest and then stand up and sit down as many times as possible within 30 seconds. The number of full stands completed is recorded. This test assesses functional lower limb muscle strength and core stability. An increase in the number of repetitions indicates an improvement in functional strength.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Result] Seckinogullari B, Balkan AF, Cakmakli GY, Aksoy S, Elibol B. Acute effects of lumbosacral mobilization on balance and functional activities in idiopathic Parkinson's disease:A randomised controlled trial. Neurol Res. 2023 Aug;45(8):745-752. doi: 10.1080/01616412.2023.2203613. Epub 2023 Apr 17. PMID 37068206
- [Result] Yang WC, Hsu WL, Wu RM, Lu TW, Lin KH. Motion analysis of axial rotation and gait stability during turning in people with Parkinson's disease. Gait Posture. 2016 Feb;44:83-8. doi: 10.1016/j.gaitpost.2015.10.023. Epub 2015 Nov 9. PMID 27004637
- [Result] Van Emmerik RE, Wagenaar RC, Winogrodzka A, Wolters EC. Identification of axial rigidity during locomotion in Parkinson disease. Arch Phys Med Rehabil. 1999 Feb;80(2):186-91. doi: 10.1016/s0003-9993(99)90119-3. PMID 10025495